CLINICAL TRIAL: NCT03945942
Title: Influence of Hyperbilirubinaemia on Foresight and INVOS Oximetry Values in Pediatric Hepatic Transplantation
Brief Title: Influence of Hyperbilirubinaemia on Two Different Near Infrared Spectroscopy Devices
Acronym: NIRS_GREFFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018/07NOV/413
Record Dates: First submitted 2019-03-04; First posted 2019-05-10 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Liver Transplant; Complications
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric liver transplant patients (Other): Using somatic and cerebral Near infrared spectroscopy devices
  Interventions: Device: Near infrared spectroscopy with INVOS device; Device: Near infrared spectroscopy with Foresight device

INTERVENTIONS:
Device: Near infrared spectroscopy with INVOS device — somatic and cerebral oximetry by INVOS in pediatric liver transplantation
Device: Near infrared spectroscopy with Foresight device — somatic and cerebral oximetry with Foresight device in pediatric liver transplantation

SUMMARY:
Protocol Near infrared spectroscopy liver transplants: comparison of two monitoring of Near infrared spectroscopy in pediatric liver transplant.

DETAILED DESCRIPTION:
Hyperbilirubinaemia may interfere with oximetry values as measured by Near Infrared Spectroscopy devices. The number of wave lengths used by different devices can influence the oximetry values in adult patients. This has never been demonstrated in children with hyperbilirubinaemia scheduled for elective liver transplantation.The study will compare cerebral and somatic oximetry values measured by two different Near infrared spectroscopy devices (FORESIGHT and INVOS) and analyse the influence of bilirubin levels on these differences.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients 0 to 18 years, with a liver transplant with living donor program of our institution
* Free, informed and written consent signed by the investigator or employees and by the legal guardians of minor patients in the days preceding the procedure

Exclusion Criteria:

* refusal of the patient or his parents to consent
* known brain or Neurological pathology

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
influence of chromophores such as bilirubin on oximetry values provided by two different devices | From Day 0 of surgery until arrival at pediatric intensive care unit (up to 12 hours)
  measure of oximetry values by two different devices at different time points in function of serum bilirubin levels

CONTACTS AND LOCATIONS:
Overall Officials: Natalia MAGASICH-AIROLA, MD, Principal Investigator — natalia.magasich@uclouvain.be
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No